CLINICAL TRIAL: NCT05255926
Title: An Exploratory, Open-Label, Single Center Study of CXCR4-targeted PET/CT Imaging for Evaluation of Hematological Malignancies
Brief Title: CXCR4-targeted PET/CT Imaging in Hematological Malignancies
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhongnan Hospital (Other)
Responsible Party: Principal Investigator, Yong He, Principal Investigator, Zhongnan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ZNYYHYXK0002
Record Dates: First submitted 2022-01-26; First posted 2022-02-25 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: CXCR4; PET/CT; Hematological Malignancy
MeSH Terms: conditions — Hematologic Neoplasms | interventions — 68Ga-pentixafor; Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 68Ga-pentixafor and 18F-FDG PET/CT (Experimental): Patients with a high clinical suspicion of, or confirmed newly diagnosed or relapsed hematological malignancies will be recruited. All enrolled patients will undergo both 68Ga-pentixafor and 18F-FDG PET/CT imaging within two weeks.
  Interventions: Drug: 68Ga-pentixafor; Device: PET/CT

INTERVENTIONS:
Drug: 68Ga-pentixafor — All participants undergo intravenous administration of 68Ga-pentixafor (1.85-3.71 MBq/kg body weight).
Device: PET/CT — PET/CT imaging is performed 1 h after intravenous injection of 68Ga-pentixafor.
  Other Names: Positron Emission Tomography/Computed Tomography

SUMMARY:
Hematological malignancies continue to pose significant clinical challenges due to their high incidence, heterogeneous biology, and substantial mortality. Although 18F-FDG PET/CT remains the most commonly used molecular imaging modality, its limited specificity can result in false-positive or false-negative findings, especially in indolent or low-metabolism subtypes, thereby hampering accurate diagnosis, staging, and therapeutic evaluation. C-X-C chemokine receptor type 4 (CXCR4) is frequently overexpressed in a broad spectrum of hematologic malignancies and correlates with aggressive disease and unfavorable outcomes. CXCR4-targeted molecular imaging using ^68Ga-pentixafor PET/CT has shown promise for improved disease characterization. This prospective study aims to systematically compare 68Ga-pentixafor PET/CT with 18F-FDG PET/CT in terms of diagnostic performance, staging accuracy, risk stratification, and prognostic relevance in patients with hematological malignancies. Furthermore, the study will incorporate artificial intelligence-based image analysis to enhance lesion detection, automate quantitative assessments, and support personalized clinical decision-making.

DETAILED DESCRIPTION:
Hematological malignancies encompass a heterogeneous group of neoplasms originating from the bone marrow and lymphatic system. Despite advances in therapeutic strategies, the prognosis for many subtypes remains suboptimal, and accurate initial evaluation is critical for appropriate treatment planning. ^18F-FDG PET/CT is routinely used for functional imaging in these patients; however, its diagnostic utility is limited by variable glucose metabolism across disease subtypes and inflammatory uptake, which can lead to misclassification.

CXCR4, a chemokine receptor involved in tumor proliferation, invasion, and microenvironmental interactions, is overexpressed in numerous hematologic malignancies and has emerged as a molecular target for both imaging and therapy. 68Ga-pentixafor, a CXCR4-targeted PET radiotracer, has demonstrated superior lesion detection in preliminary studies, particularly in diseases with low 18F-FDG avidity.

This prospective study will investigate the clinical utility of 68Ga-pentixafor PET/CT in patients with newly diagnosed or relapsed hematological malignancies. Comparative analyses with 18F-FDG PET/CT will be performed to assess concordance, staging accuracy, and association with known risk stratification systems. Longitudinal follow-up will be conducted to evaluate the prognostic relevance of imaging findings.

In parallel, the study will explore the application of artificial intelligence (AI) techniques, including deep learning-based image segmentation and radiomic feature extraction, to enhance diagnostic precision and support risk-adapted management strategies. AI-driven models will be developed and validated to predict disease burden, progression, and survival, thereby contributing to personalized medicine in hematologic oncology.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteer to participate and sign an informed consent form;
2. 18 ≤ Age ≤ 90 years;
3. Patients with highly suspected, or newly diagnosed, or relapsed hematological malignancies;
4. Willing and able to follow schedule visits, treatment plans and laboratory tests.

Exclusion Criteria:

1. pregnancy or breastfeeding;
2. Allergic to CXCR4-targeted tracers or excipients;
3. Fasting blood glucose level exceeded 11.0 mmol/L prior to injection of 18F-FDG;
4. Those who cannot complete PET/CT scan, including inability to keep supine, claustrophobia, radiation phobia, etc.;
5. Researchers think it is inappropriate to participate in this clinical trial for patients with poor compliance or other unsuitable factors.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Accuracy of 68Ga-pentixafor PET/CT Compared to 18F-FDG PET/CT in Hematological Malignancies | Two years
  To assess and compare the diagnostic accuracy of 68Ga-pentixafor PET/CT and 18F-FDG PET/CT in patients with newly diagnosed, relapsed, or highly suspected hematological malignancies. Accuracy will be evaluated using a composite reference standard, including histopathological confirmation, clinical follow-up, and additional imaging findings.
Concordance of [⁶⁸Ga]Ga-pentixafor PET/CT with Standard Clinical Staging Systems | Two years
  To evaluate the concordance between [⁶⁸Ga]Ga-pentixafor PET/CT-based staging and conventional clinical staging systems (e.g., Ann Arbor, Durie-Salmon PLUS, R-ISS/R2-ISS) in patients with hematological malignancies. Concordance will be measured using Cohen's kappa statistic (κ).
Predictive Value of [⁶⁸Ga]Ga-pentixafor PET/CT Parameters for Progression-Free Survival | Four years
  To assess whether imaging biomarkers from [⁶⁸Ga]Ga-pentixafor PET/CT, such as SUVmax or total lesion CXCR4 uptake, predict progression-free survival (PFS) in patients with hematological malignancies. Comparison will be made with [¹⁸F]FDG PET/CT-derived parameters.
Predictive Value of [⁶⁸Ga]Ga-pentixafor PET/CT Parameters for Overall Survival | Four years
  To evaluate whether [⁶⁸Ga]Ga-pentixafor PET/CT-based biomarkers can predict overall survival in patients with hematological malignancies, compared with [¹⁸F]FDG PET/CT.
Dice Similarity Coefficient (DSC) for AI-based lesion segmentation | Two years
  Evaluation of the overlap between artificial intelligence-generated lesion segmentations and expert manual annotations on PET/CT images using the Dice similarity coefficient (DSC).

SECONDARY OUTCOMES:
Correlation Between CXCR4 Expression and [⁶⁸Ga]Ga-pentixafor PET/CT Parameters | Two years
  To assess the correlation between CXCR4 expression levels in biopsy samples and semiquantitative parameters from [⁶⁸Ga]Ga-pentixafor PET/CT (e.g., SUVmax).
Correlation between del(17p) status and TLU on [68Ga]Ga-pentixafor PET/CT | Two years
  To assess the correlation between the presence or absence of del(17p), as identified by fluorescence in situ hybridization (FISH), and total lesion uptake (TLU) on [68Ga]Ga-pentixafor PET/CT at baseline. The degree of correlation will be measured using the Spearman correlation coefficient (rho), a unitless value ranging from -1 to +1.
Radiogenomic Model for Risk Prediction Using AI | Two years
  To develop and validate an AI-based radiogenomic model integrating PET imaging features and genomic data to predict disease aggressiveness in patients with hematological malignancies.

CONTACTS AND LOCATIONS:
Overall Officials: Yong He, MD, PhD, Principal Investigator — Zhongnan Hospital
Locations (1):
- Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Herrmann K, Lapa C, Wester HJ, Schottelius M, Schiepers C, Eberlein U, Bluemel C, Keller U, Knop S, Kropf S, Schirbel A, Buck AK, Lassmann M. Biodistribution and radiation dosimetry for the chemokine receptor CXCR4-targeting probe 68Ga-pentixafor. J Nucl Med. 2015 Mar;56(3):410-6. doi: 10.2967/jnumed.114.151647. Epub 2015 Feb 19. PMID 25698782
- [Background] Pan Q, Cao X, Luo Y, Li J, Feng J, Li F. Chemokine receptor-4 targeted PET/CT with 68Ga-Pentixafor in assessment of newly diagnosed multiple myeloma: comparison to 18F-FDG PET/CT. Eur J Nucl Med Mol Imaging. 2020 Mar;47(3):537-546. doi: 10.1007/s00259-019-04605-z. Epub 2019 Nov 27. PMID 31776631
- [Background] Duell J, Krummenast F, Schirbel A, Klassen P, Samnick S, Rauert-Wunderlich H, Rasche L, Buck AK, Wester HJ, Rosenwald A, Einsele H, Topp MS, Lapa C, Kircher M. Improved Primary Staging of Marginal-Zone Lymphoma by Addition of CXCR4-Directed PET/CT. J Nucl Med. 2021 Oct;62(10):1415-1421. doi: 10.2967/jnumed.120.257279. Epub 2021 Feb 12. PMID 33579803